CLINICAL TRIAL: NCT04310280
Title: Effects of Local Insulin on Wound Angiogenesis and Fibroplasia in Varicose Ulcers
Brief Title: Effects of Local Insulin on Varicose Ulcers for Wound Healing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, MARIO AURELIO MARTÍNEZ-JIMÉNEZ, Professor, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-17
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Chronic Venous Disease; Varicose Ulcer; Wound Healing; Insulin; Angiogenesis
Keywords: Varicose Ulcer; Wound Healing; Insulin; Angiogenesis
MeSH Terms: conditions — Varicose Ulcer; Insulin Resistance | interventions — Insulin Glargine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel assignment Randomized split-plot design
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Double Blind (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical insulin glargine (Experimental): The wound surface is treated locally with glargine insulin injected sub-dermal in a daily matter for 7 days. Allocation is randomized.
  Interventions: Drug: Insulin Glargine
- 0.9% saline solution (Placebo Comparator): The wound surface is treated with conventional wound care in a daily matter for 7 days. Allocation is randomized.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Insulin Glargine — Half of the wound surface is injected daily with topical glargine insulin
  Arms: Topical insulin glargine
Drug: Saline — Half of the wound surface is injected daily with topical saline solution
  Arms: 0.9% saline solution

SUMMARY:
A randomized, split-plot, double-blind, placebo-controlled trial. The varicose ulcer is divided into two (side A and B). Half of the wound's surface is treated locally with insulin (Glargine) applied at an approx depth of 3-4 mm. Treatment with insulin is administered for 7 days. Biopsy specimens of the two sides are obtained on days 0 and 7. A thermographic photograph of the wound is taken at days 0 and 7. The number of blood vessels and fibroplasia is evaluated as the main outcome.

DETAILED DESCRIPTION:
A randomized, split-plot, double-blind, placebo-controlled trial. Chronic Varicose Ulcers measuring more than 4 cm in any of its dimensions, and that comply with candidate criteria are included in the present study. A split-mouth model is used.

The ulcer is divided into two (sides A and B). The side in which treatment is applied is randomized. Half of the wound's surface is treated locally with insulin (Glargine) applied at an approx depth of 3-4 mm. Both halves are covered with dressings and compression therapy is applied. Treatment with insulin is administered for 7 days. Biopsy specimens of the two sides are obtained on days 0 and 7. A thermographic photograph of the wound is taken at days 0 and 7, as control of the local temperature of the wound. This is to asses the process of healing and to correlate with our outcome measures. The number of blood vessels will be evaluated as the main outcome. Fibroplasia and thermal asymmetry between wound sides will be evaluated as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Presence of varicose ulcer in lower extremities with a size greater than 25 cm2
* Absence of infection

Exclusion Criteria:

* Presence of diabetes or glycated hemoglobin >6.5%
* Comorbidities that affect wound healing
* Malnutrition
* Active smoking

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Final angiogenesis | Day 7
  Number of blood vessels in a skin biopsy

SECONDARY OUTCOMES:
Fibroplasia | Day 7
  Percentage of fibrous tissue in a skin biopsy
Thermal asymmetry | Day 7
  Difference between the temperature of the wound and the surrounding healthy tissue
Hypoglycaemia | Day 7
  Presence of capillary blood glucose of <60 mg/dl or clinical symptoms of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Ramirez-GarciaLuna, MD, PhD, Study Chair — Universidad Autonoma de San Luis Potosí
Locations (1):
- Mario Aurelio Martínez-Jiménez, San Luis Potosí City, San Luis Potosí, Mexico

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be available upon request after the publication of results.

REFERENCES:
- [Result] Martinez-Jimenez MA, Valadez-Castillo FJ, Aguilar-Garcia J, Ramirez-GarciaLuna JL, Gaitan-Gaona FI, Pierdant-Perez M, Valdes-Rodriguez R, Sanchez-Aguilar JM. Effects of Local Use of Insulin on Wound Healing in Non-diabetic Patients. Plast Surg (Oakv). 2018 May;26(2):75-79. doi: 10.1177/2292550317740688. Epub 2017 Nov 22. PMID 29845043
- [Result] Martinez-Jimenez MA, Aguilar-Garcia J, Valdes-Rodriguez R, Metlich-Medlich MA, Dietsch LJP, Gaitan-Gaona FI, Kolosovas-Machuca ES, Gonzalez FJ, Sanchez-Aguilar JM. Local use of insulin in wounds of diabetic patients: higher temperature, fibrosis, and angiogenesis. Plast Reconstr Surg. 2013 Dec;132(6):1015e-1019e. doi: 10.1097/PRS.0b013e3182a806f0. PMID 24281606
- [Derived] Martinez-Jimenez MA, Kolosovas-Machuca S, Alcocer F, Ortiz-Dosal LC, Gonzalez-Grijalva MC, Delsol-Revuelta GA, Gaitan-Gaona FI, Valadez-Castillo FJ, Ramirez-GarciaLuna JL. A Randomized Controlled Trial on the Effect of Local Insulin Glargine on Venous Ulcer Healing. J Surg Res. 2022 Nov;279:657-665. doi: 10.1016/j.jss.2022.06.070. Epub 2022 Aug 3. PMID 35932720